CLINICAL TRIAL: NCT07205380
Title: GallRiks ERC Anesthesia Study
Status: Completed | Type: Observational
Sponsor: Karolinska Institutet (Other)
Responsible Party: Principal Investigator, Gabriel Sandblom, Associate Professor, Karolinska Institutet
Other Study IDs: GallRiks ERC anesthesia study
Record Dates: First submitted 2025-09-19; First posted 2025-10-03 (Actual); Last update posted 2025-10-03 (Actual); Status verified 2025-09

CONDITIONS: Gallstone Disease
Keywords: gallstone; ERCP; Anesthesia
MeSH Terms: conditions — Cholelithiasis; Gallstones

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Swedish National Register for Gallstone Surgery and ERCP: Interventions for gallstones registered in Sweden
  Interventions: Procedure: Endoscopic Retrograde Cholangiopancreaticography

INTERVENTIONS:
Procedure: Endoscopic Retrograde Cholangiopancreaticography — Anaesthesia or sedation during ERCP for common bile duct stones

SUMMARY:
Endoscopic retrograde cholangiopancreatography (ERCP) for common bile duct stones (CBDS) removal can be performed under varying levels of sedation. Deeper sedation has been associated with more successful cannulation, but little is known about the efficacy of ERCP measured as rate of retained CBDS depending on the level of sedation.

In this population-based, cohort study, using prospectively assembled register data from 121 252 ERCP procedures, adjusted odds ratio (OR) of retained CBDS 12 months after CBDS removal are analysed. Retained CBDS are defined as a repeated ERCP where CBDS are found.

ELIGIBILITY:
Inclusion Criteria:

* ERCP performed for common bile duct stones

Exclusion Criteria:

* Suspicion of bile duct tumour
* ERCP performed during the seanse as a cholecystectomy
* Patients having undergone ERCP previously

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients undergoing ERCP for common bile duct stones
Sampling Method: Non-Probability Sample
Enrollment: 121252 (Actual)
Dates: Start 2007-01-01 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
Incidence of ERCP for retained stones performed after the primary ERCP. | 12 months
  Retained common bile duct stones necessitating repeated ERCP within 12 months after the first ERCP

IPD SHARING:
Plan to Share IPD: Yes
Pseudonymized data from the study are available on request from Gabriel Sandblom
Supporting Information: Study Protocol, SAP
Time Frame: 2025-09-18 - 2025-12-31
Access Criteria: Researchers presenting their position and reason for accessing the IPD.